CLINICAL TRIAL: NCT04275752
Title: Examining the Preliminary Efficacy, Feasibility, and Acceptability of an Exercise Intervention on Frailty After Kidney Transplantation
Brief Title: Exercise Intervention on Frailty After Kidney Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Original funding for this study changed and it is no longer being pursued
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth C. Lorenz, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-008545; K23DK123313-01 (NIH)
Record Dates: First submitted 2020-02-13; First posted 2020-02-19 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): Subjects will receive no formal exercise recommendations
- Exercise Intervention Group (Experimental): Subjects will complete an exercise program
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Exercise Program — Perform endurance (treadmill or cycle ergometer), strength (weight resistance), and flexibility training twice a week for a period of one hour per session, for a total of 16 sessions.
  Arms: Exercise Intervention Group

SUMMARY:
Researchers are trying to determine if exercise will improve health and strength in kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years who have received a KT and have a functioning allograft

Exclusion Criteria:

* Neuropsychiatric condition causing patient to be unable to provide consent
* Recipient of a combined organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in frailty status | Two months
  Frailty will be determined by Frailty Phenotype (FP) or Short Physical Performance Battery (SPPB) scores. FP is determined by the presence of 3 or more of the following: slowness (measured by gait speed), exhaustion (measured via self-report), weakness (measured by hand grip strength), low physical activity level (measured via self-report), and wasting (measured via self-report or by tracking changes in weight). The SPPB consists of a gait speed test, balance testing, and repeated chair stands. A score less than or equal to 10 will be considered frail.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lorenz, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials